CLINICAL TRIAL: NCT05638529
Title: Dual Versus Single Trigger in IVF Patients at High Risk of Ovarian Hyper Stimulation Syndrome: a Randomized, Double-blinded, Controlled Trial.
Brief Title: Dual Trigger" in IVF Patients at High Risk of Ovarian Hyper Stimulation Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Miguel Angel Russo, Physician, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-0302-A
Record Dates: First submitted 2022-11-23; First posted 2022-12-06 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Ovarian Hyperstimulation Syndrome; Infertility, Female
Keywords: oocyte Maturity; Dual Trigger; Infertility, Female
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome; Infertility, Female | interventions — Chorionic Gonadotropin; Thyrotropin Alfa; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm- Group A (Experimental): A subcutaneous injection of a GnRH agonist (Suprefact 0.5 mg) and a separate intramuscular injection of hCG (Pregnyl 1,500 IU).
  Interventions: Drug: Pregnyl (1,500) IU
- Control Arm- Group B (Placebo Comparator): A subcutaneous injection of a GnRH agonist (Suprefact 0.5 mg) and a separate intramuscular injection of normal saline (1.5 mL) (sham-placebo).
  Interventions: Drug: 1.5 mL of normal saline

INTERVENTIONS:
Drug: Pregnyl (1,500) IU — Patients will self-administer a subcutaneous injection of a GnRH agonist (Suprefact 0.5 mg) and a separate intramuscular injection of hCG (Pregnyl 1,500 IU) on their assigned trigger day.
  Other Names: Hcg
  Arms: Treatment Arm- Group A
Drug: 1.5 mL of normal saline — Patients will self-administer a subcutaneous injection of a GnRH agonist (Suprefact 0.5 mg) and a separate intramuscular injection of normal saline (1.5 mL - sham placebo) on their assigned trigger day.
  Other Names: Normal Saline
  Arms: Control Arm- Group B

SUMMARY:
The present study aims to evaluate whether the use of a "dual trigger" can improve IVF outcomes, compared to GnRH agonist (GnRH-a) alone, in patients at high risk of OHSS undergoing a freeze-all cycle. By examining freeze-all cycles with frozen embryo transfer(s) (FET) only, we eliminate the potential confounding issue of inadequate luteal support to the endometrium and focus primarily on the effect of a "dual trigger" on oocyte quality and embryo potential.

To our best knowledge, there have been no randomized, controlled trials conducted to address this hypothesis.

DETAILED DESCRIPTION:
While the use of GnRH-a trigger has nearly eliminated the risk of OHSS, several studies have shown that this strategy may be associated with poorer IVF outcomes after a fresh embryo transfer (Engmann et al., 2008; Galindo et al., 2009; Melo et al., 2017; Sismanoglu et al., 2009; Youssef et al., 2014). These findings may be partly explained by an inadequate LH surge, following a GnRH-a trigger, and raises two separate concerns. The first concern is whether an inadequate LH surge can have an detrimental effect on luteal support following a fresh embryo transfer. The corpus luteum requires constant LH stimulation, during implantation and early gestation, in order to optimize endometrial receptivity via the production of progesterone. The second concern is whether a suboptimal LH surge can reduce the number or quality of mature oocytes retrieved during a treatment cycle. Immature oocytes will not fertilize invitro and, therefore, can decrease a woman's overall success rate with IVF. Based on this second premise, another strategy was developed whereby a "dual trigger", using a combination of a GnRH-a and a lower dose of hCG (1,500 IU), is used to help maximize the number of "mature eggs" retrieved during an IVF cycle without increasing the risk of OHSS. Two recent retrospective studies have evaluated the administration of a "dual trigger" with GnRH agonist in combination with low-dose hCG (1,000 IU), compared to GnRH agonist alone (O'Neill et al., 2016; Griffin et al., 2012). Both studies revealed a significant improvement in the number of mature oocytes retrieved between treatment and controls (Griffin et al., 2012). While these findings are promising, it is important to note that oocyte maturity does not equate to embryo potential. Therefore, whether the use of a "dual trigger" improves embryo development and competency, thus increasing a patient's success rate, remains to be determined.

ELIGIBILITY:
Inclusion Criteria:

* They are between the ages of 18 and 40.
* They are undergoing IVF treatment with a GnRH antagonist protocol.
* During their current treatment cycle, they have at least one of the following risk factors for OHSS:

  * Greater or equal to 13 follicles measuring at least 11 mm on the day of trigger.
  * Serum estradiol levels greater or equal to 15,000 pmol/L on the day of trigger.

Exclusion Criteria:

* They are using a GnRH agonist protocol (which is a contraindication to using a GnRH agonist trigger).
* They are planning on using a "dual trigger" (based on poor outcomes in a previous IVF cycle using a GnRH agonist trigger).
* They have a low ovarian reserve (AFC < 7 follicles or AMH < 10 pmol/L).
* They have had a previous failed GnRH agonist trigger.
* They have a known diagnosis of hypogonadotropic hypogonadism.
* They have had a previous adverse or allergic reaction to GnRH agonist in the past.
* They are using surgically retrieved sperm.
* They are undergoing treatment for fertility preservation (oncofertility patients).
* They have a history of recurrent implantation failure (defined as no clinical pregnancy after transfer of > 4 good-quality embryos).
* They have any congenital or acquire uterine anomalies distorting the uterine cavity.
* If serum estradiol levels are equal or exceed 28,000 pmol/L on the day of trigger

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Total number of Day 5 embryos | after 5 days of oocyte fertilization
  Total number of "good quality" Day 5 embryos available for cryopreservation.

SECONDARY OUTCOMES:
Total number of oocytes retrieved per cycle. | within 1-2 days of oocyte retrieval
Total number of mature oocytes (MII) retrieve per IVF/ICSI cycle. | 2-3 days after oocyte retrieval
Total number of fertilized zygotes. | 3-5 days after the egg retrieval
Fertilization rate | 3-5 days after the egg retrieval
  Number of 2PN zygote(s) divided by the number of mature oocyte(s) fertilized per IVF/ICSI cycle OR Number of 2PN zygote(s) divided by the number of oocytes incubated with at least 10,000 sperm per IVF cycle.
Total number of Day 3 embryos. | 3 days after the fertilization of oocyte
Pregnancy Rate | Upto 13 weeks after the embryo transfer
  A serum b-hCG > 5 mIU/mL per transfer
Clinical pregnancy rate | Upto 13 weeks after the embryo transfer
  Number of gestational sac(s) with a positive fetal heart per transfer.
Implantation rate | 3-4 weeks after implantation of embryos
  Number of gestational sac(s) divided by the number of embryo(s) transferred per FET.
Miscarriage rate | Within 20 weeks from the date of the clinical intrauterine pregnancy confirmation ultrasount
  The number of spontaneous pregnancy losses before 20 weeks gestation divided by the number of clinical pregnancies
Live birth rate | Per embryo(s) transferred during the study period and follow-up for up to 10 months after last transfer.]
  The number of live born neonates over 24 weeks gestation divided by the number of clinical pregnancies
Incidence of moderate to critical OHSS | Upto 2 weeks from the date of intervention
  Based on the classification criteria by Mathur et al. (2007).

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Russo, MD, Principal Investigator — Mount Sinai Hospital, Canada
Locations (1):
- Mount Sinai Hospital, Fertility Clinic, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Corbett S, Shmorgun D, Claman P; REPRODUCTIVE ENDOCRINOLOGY INFERTILITY COMMITTEE; SPECIAL CONTRIBUTOR. The prevention of ovarian hyperstimulation syndrome. J Obstet Gynaecol Can. 2014 Nov;36(11):1024-1033. doi: 10.1016/S1701-2163(15)30417-5. English, French. PMID 25574681
- [Background] Rotterdam ESHRE/ASRM-Sponsored PCOS Consensus Workshop Group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome. Fertil Steril. 2004 Jan;81(1):19-25. doi: 10.1016/j.fertnstert.2003.10.004. PMID 14711538
- [Background] Ferraretti AP, Gianaroli L, Magli C, Fortini D, Selman HA, Feliciani E. Elective cryopreservation of all pronucleate embryos in women at risk of ovarian hyperstimulation syndrome: efficiency and safety. Hum Reprod. 1999 Jun;14(6):1457-60. doi: 10.1093/humrep/14.6.1457. PMID 10357958
- [Background] Galindo A, Bodri D, Guillen JJ, Colodron M, Vernaeve V, Coll O. Triggering with HCG or GnRH agonist in GnRH antagonist treated oocyte donation cycles: a randomised clinical trial. Gynecol Endocrinol. 2009 Jan;25(1):60-6. doi: 10.1080/09513590802404013. PMID 19165664
- [Background] Griffin D, Benadiva C, Kummer N, Budinetz T, Nulsen J, Engmann L. Dual trigger of oocyte maturation with gonadotropin-releasing hormone agonist and low-dose human chorionic gonadotropin to optimize live birth rates in high responders. Fertil Steril. 2012 Jun;97(6):1316-20. doi: 10.1016/j.fertnstert.2012.03.015. Epub 2012 Apr 3. PMID 22480822
- [Background] Huang CY, Shieh ML, Li HY. The benefit of individualized low-dose hCG support for high responders in GnRHa-triggered IVF/ICSI cycles. J Chin Med Assoc. 2016 Jul;79(7):387-93. doi: 10.1016/j.jcma.2016.02.006. Epub 2016 May 1. PMID 27147462
- [Background] Lin H, Wang W, Li Y, Chen X, Yang D, Zhang Q. Triggering final oocyte maturation with reduced doses of hCG in IVF/ICSI: a prospective, randomized and controlled study. Eur J Obstet Gynecol Reprod Biol. 2011 Nov;159(1):143-7. doi: 10.1016/j.ejogrb.2011.07.009. Epub 2011 Aug 6. PMID 21824709
- [Background] Ludwig M, Doody KJ, Doody KM. Use of recombinant human chorionic gonadotropin in ovulation induction. Fertil Steril. 2003 May;79(5):1051-9. doi: 10.1016/s0015-0282(03)00173-0. PMID 12738494
- [Background] McClure N, Healy DL, Rogers PA, Sullivan J, Beaton L, Haning RV Jr, Connolly DT, Robertson DM. Vascular endothelial growth factor as capillary permeability agent in ovarian hyperstimulation syndrome. Lancet. 1994 Jul 23;344(8917):235-6. doi: 10.1016/s0140-6736(94)93001-5. PMID 7913160
- [Background] Melo M, Busso CE, Bellver J, Alama P, Garrido N, Meseguer M, Pellicer A, Remohi J. GnRH agonist versus recombinant HCG in an oocyte donation programme: a randomized, prospective, controlled, assessor-blind study. Reprod Biomed Online. 2009 Oct;19(4):486-92. doi: 10.1016/j.rbmo.2009.06.001. PMID 19909588
- [Background] Nargund G, Hutchison L, Scaramuzzi R, Campbell S. Low-dose HCG is useful in preventing OHSS in high-risk women without adversely affecting the outcome of IVF cycles. Reprod Biomed Online. 2007 Jun;14(6):682-5. doi: 10.1016/s1472-6483(10)60668-2. PMID 17579978
- [Background] Neulen J, Yan Z, Raczek S, Weindel K, Keck C, Weich HA, Marme D, Breckwoldt M. Human chorionic gonadotropin-dependent expression of vascular endothelial growth factor/vascular permeability factor in human granulosa cells: importance in ovarian hyperstimulation syndrome. J Clin Endocrinol Metab. 1995 Jun;80(6):1967-71. doi: 10.1210/jcem.80.6.7775647.
- [Background] O'Neill KE, Senapati S, Maina I, Gracia C, Dokras A. GnRH agonist with low-dose hCG (dual trigger) is associated with higher risk of severe ovarian hyperstimulation syndrome compared to GnRH agonist alone. J Assist Reprod Genet. 2016 Sep;33(9):1175-84. doi: 10.1007/s10815-016-0755-8. Epub 2016 Jun 27. PMID 27349252
- [Background] Oktay K, Turkcuoglu I, Rodriguez-Wallberg KA. GnRH agonist trigger for women with breast cancer undergoing fertility preservation by aromatase inhibitor/FSH stimulation. Reprod Biomed Online. 2010 Jun;20(6):783-8. doi: 10.1016/j.rbmo.2010.03.004. Epub 2010 Mar 6. PMID 20382080
- [Background] Orvieto R, Rabinson J, Meltzer S, Zohav E, Anteby E, Homburg R. Substituting HCG with GnRH agonist to trigger final follicular maturation--a retrospective comparison of three different ovarian stimulation protocols. Reprod Biomed Online. 2006 Aug;13(2):198-201. doi: 10.1016/s1472-6483(10)60615-3. PMID 16895632
- [Background] Papanikolaou EG, Pozzobon C, Kolibianakis EM, Camus M, Tournaye H, Fatemi HM, Van Steirteghem A, Devroey P. Incidence and prediction of ovarian hyperstimulation syndrome in women undergoing gonadotropin-releasing hormone antagonist in vitro fertilization cycles. Fertil Steril. 2006 Jan;85(1):112-20. doi: 10.1016/j.fertnstert.2005.07.1292. PMID 16412740
- [Background] Pellicer A, Albert C, Mercader A, Bonilla-Musoles F, Remohi J, Simon C. The pathogenesis of ovarian hyperstimulation syndrome: in vivo studies investigating the role of interleukin-1beta, interleukin-6, and vascular endothelial growth factor. Fertil Steril. 1999 Mar;71(3):482-9. doi: 10.1016/s0015-0282(98)00484-1. PMID 10065786
- [Background] Practice Committee of the American Society for Reproductive Medicine. Electronic address: ASRM@asrm.org; Practice Committee of the American Society for Reproductive Medicine. Prevention and treatment of moderate and severe ovarian hyperstimulation syndrome: a guideline. Fertil Steril. 2016 Dec;106(7):1634-1647. doi: 10.1016/j.fertnstert.2016.08.048. Epub 2016 Sep 24. PMID 27678032
- [Background] Revelli A, Carosso A, Grassi G, Gennarelli G, Canosa S, Benedetto C. Empty follicle syndrome revisited: definition, incidence, aetiology, early diagnosis and treatment. Reprod Biomed Online. 2017 Aug;35(2):132-138. doi: 10.1016/j.rbmo.2017.04.012. Epub 2017 May 23. PMID 28596003
- [Background] Schmidt DW, Maier DB, Nulsen JC, Benadiva CA. Reducing the dose of human chorionic gonadotropin in high responders does not affect the outcomes of in vitro fertilization. Fertil Steril. 2004 Oct;82(4):841-6. doi: 10.1016/j.fertnstert.2004.03.055. PMID 15482757
- [Background] Shaker AG, Zosmer A, Dean N, Bekir JS, Jacobs HS, Tan SL. Comparison of intravenous albumin and transfer of fresh embryos with cryopreservation of all embryos for subsequent transfer in prevention of ovarian hyperstimulation syndrome. Fertil Steril. 1996 May;65(5):992-6. doi: 10.1016/s0015-0282(16)58275-2. PMID 8612863
- [Background] Shapiro BS, Daneshmand ST, Garner FC, Aguirre M, Hudson C. Comparison of "triggers" using leuprolide acetate alone or in combination with low-dose human chorionic gonadotropin. Fertil Steril. 2011 Jun 30;95(8):2715-7. doi: 10.1016/j.fertnstert.2011.03.109. Epub 2011 May 7. PMID 21550042
- [Background] Youssef MA, Van der Veen F, Al-Inany HG, Mochtar MH, Griesinger G, Nagi Mohesen M, Aboulfoutouh I, van Wely M. Gonadotropin-releasing hormone agonist versus HCG for oocyte triggering in antagonist-assisted reproductive technology. Cochrane Database Syst Rev. 2014 Oct 31;2014(10):CD008046. doi: 10.1002/14651858.CD008046.pub4. PMID 25358904
- [Background] Sismanoglu A, Tekin HI, Erden HF, Ciray NH, Ulug U, Bahceci M. Ovulation triggering with GnRH agonist vs. hCG in the same egg donor population undergoing donor oocyte cycles with GnRH antagonist: a prospective randomized cross-over trial. J Assist Reprod Genet. 2009 May;26(5):251-6. doi: 10.1007/s10815-009-9326-6. Epub 2009 Jul 23. PMID 19629674
- [Background] Werner, M. D., Forman, E. J., Hong, K. H., Franasiak, J. M., Neal, S. A., & Scott, R. T. (2014). Dual trigger with GnRH agonist (GnRHa) and varying doses of hCG increases the blastulation rate amongst high responders. Fertility and Sterility, 102(3), e220
- [Background] Angelo, D. A., & Nn, A. (2012). Embryo freezing for preventing ovarian hyperstimulation syndrome (Review) SUMMARY OF FINDINGS FOR THE MAIN COMPARISON, (3).
- [Background] Shaltout, A., Eid, M., & Shohayeb, A. (2006). Does triggering ovulation by 5000 IU of uhCG affect ICSI outcome? Middle East Fertility Society Journal, 11: 99-103.
- [Background] Gardner DK, Schoolcraft WB. In vitro culture of human blastocyst. In: Janson R, Mortimer D, editors. Towards Reproductive Certainty: Infertility and Genetics Beyond 1999. Carnforth: Parthenon Press; 1999. p. 378-88.